CLINICAL TRIAL: NCT03894345
Title: Open Label 8-Week Study of Prazosin Use in Adults With Anxiety Disorders
Brief Title: Prazosin Use in Adults With Anxiety Disorders
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS21444 (B2018:002) PRA2051N
Record Dates: First submitted 2019-02-14; First posted 2019-03-28 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Anxiety; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Prazosin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label treatment with Prazosin (Experimental): Week 1 Day 1-3: 0.5 mg at bedtime Day 4-7: 1.0 mg at bedtime Week 2 Day 8-10: 2.0 mg at bedtime Day 11-14: 4.0 mg at bedtime Week 3 2 mg in the morning, 4 mg at bedtime Week 4 4 mg in the morning, 4 mg at bedtime Week 5 4 mg in the morning, 6 mg at bedtime Week 6 4 mg in the morning, 8 mg at bedtime
  Dosage of Prazosin will be titrated at the discretion of the study physician.
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Prazosin — Competitive alpha-1 adrenergic receptor blocker which has been used to treat PTSD and Benign Prostatic Hypertrophy
  Other Names: Minipress

SUMMARY:
Prazosin has shown effectiveness in treating Post-Traumatic Stress Disorder through improving sleep quality and global functioning. Given the significant evidence for its utility in treating PTSD, in combination with the fact that many anxiety symptoms overlap with PTSD (e.g.insomnia, hyperarousal, and irritability), it is essential to evaluate its potential effectiveness in treating symptoms of other anxiety disorder and patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Existing Diagnosis of any anxiety disorder according to DSM-5 criteria (i.e. GAD, Panic Disorder, Agoraphobia, Social Phobia or Specific phobias)
2. Newly diagnosed patients or patients who are either resistant or not adherent to their current treatment are eligible to be enrolled in the study.
3. If patient is on anti-hypertensive therapy, the dose of anti-hypertensive(s) must be stable for at least 4 weeks prior to the study and blood pressure must be well controlled.

Exclusion Criteria:

1. Patients with comorbid condition of psychosis, a diagnosis of PTSD, an active severe substance use disorder, or actively suicidal.
2. Patients actively enrolled in psychotherapy sessions at the time of the study.
3. Patients experiencing baseline systolic blood pressure ≤100 mmHg supine, orthostatic hypotension (a decrease in systolic blood pressure from a sitting position of 20 mmHg or more after 2 minutes standing accompanied with light-headedness), or a baseline diastolic blood pressure less than 60 mmHg.
4. Pregnant or lactating women.
5. Patients with acute medical or psychiatric conditions that require immediate hospital admission.
6. Patients with a history of allergic reaction to prazosin or any of its components.
7. Patients unable to communicate in English.
8. Patients who are scheduled to undergo cataract surgery are excluded from the study until after the surgery has been completed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Symptoms | To be completed at baseline and weekly during weeks 2,3,4,5,6,7, 8 to assess changes over the last week
  The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items, each defined by a series of, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change in Anxiety Symptoms | To be completed at baseline and weekly during weeks 2,3,4,5,6,7,8 to assess changes over the last week
  Generalized Anxiety Disorder 7 Item Scale (GAD-7) objectively determines initial symptoms severity and monitor symptom changes/effect of treatment over time. Each item is scored on a scale of "0" (not at all) to "3" (nearly every day). Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.

SECONDARY OUTCOMES:
Change in Depressive Symptoms | To be completed at baseline,weeks 2, 4 and 8 to assess changes since last previous 2 weeks
  To examine depressive symptoms following the use of prazosin as measured by the Patient Health Questionnaire (PHQ-9).Each item is scored on a scale of "0" (not at all) to "3" (nearly every day). Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Change in Level of Disability | To be completed at baseline, weeks 2, 4 and 8 to assess changes over the previous 2 weeks
  To examine levels of disability following the use of prazosin as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Change in Overall Symptom Severity | Previous 2 weeks
  To examine overall symptom severity following the use of prazosin as measured by the DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure for Adults (DSM-5).
Changes in Experienced Symptoms | Completed at Baseline, and at weeks 2, 3, 4, 5, 6, 7, 8 to assess changes over the past week
  To examine improvement in symptoms as measured by the Clinical Global Impression-Improvement Scale (CGI-I). Scale ranges from 1 (very much improved since initiation of treatment) to 7 (very much worse since initiation of treatment)
Tolerability of Medication (Heart Rate) | To be assessed at Baseline, and at weeks 2, 3, 4, 5, 6, 7, 8 to monitor changes since last visit
  To examine the overall tolerability of prazosin by recording heart rate at each visit
Tolerability of Medication (blood pressure) | To be assessed at Baseline, and at weeks 2, 3, 4, 5, 6, 7, 8
  To examine the overall tolerability of prazosin by recording blood pressure at each visit in the sitting and standing positions
Side Effects | To be assessed at Baseline, and at weeks 2, 3, 4, 5, 6, 7, 8
  To examine the overall tolerability and side effects of prazosin by recording potential adverse symptoms using a Vital Signs and Adverse Symptoms Checklist.
Change in Sleep Impairment | Will be completed by patients at baseline, weeks 2,4 and 8 to assess changes over the previous 2 weeks
  To examine sleep quality following the use of prazosin as measured by the Insomnia Severity Index (ISI).

CONTACTS AND LOCATIONS:
Overall Officials: Jitender Sareen, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba - PsycHealth - Mood and Anxiety Disorders Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Nelson CB, McGonagle KA, Edlund MJ, Frank RG, Leaf PJ. The epidemiology of co-occurring addictive and mental disorders: implications for prevention and service utilization. Am J Orthopsychiatry. 1996 Jan;66(1):17-31. doi: 10.1037/h0080151. PMID 8720638
- [Background] Bland RC, Newman SC, Orn H. Period prevalence of psychiatric disorders in Edmonton. Acta Psychiatr Scand Suppl. 1988;338:33-42. doi: 10.1111/j.1600-0447.1988.tb08545.x. PMID 3165593
- [Background] Dick CL, Bland RC, Newman SC. Epidemiology of psychiatric disorders in Edmonton. Panic disorder. Acta Psychiatr Scand Suppl. 1994;376:45-53. PMID 8178684
- [Background] Wittchen HU, Carter RM, Pfister H, Montgomery SA, Kessler RC. Disabilities and quality of life in pure and comorbid generalized anxiety disorder and major depression in a national survey. Int Clin Psychopharmacol. 2000 Nov;15(6):319-28. doi: 10.1097/00004850-200015060-00002. PMID 11110007
- [Background] Baldwin DS, Waldman S, Allgulander C. Evidence-based pharmacological treatment of generalized anxiety disorder. Int J Neuropsychopharmacol. 2011 Jun;14(5):697-710. doi: 10.1017/S1461145710001434. Epub 2011 Jan 7. PMID 21211105
- [Background] Opbroek A, Delgado PL, Laukes C, McGahuey C, Katsanis J, Moreno FA, Manber R. Emotional blunting associated with SSRI-induced sexual dysfunction. Do SSRIs inhibit emotional responses? Int J Neuropsychopharmacol. 2002 Jun;5(2):147-51. doi: 10.1017/S1461145702002870. PMID 12135539
- [Background] Birnbaum S, Gobeske KT, Auerbach J, Taylor JR, Arnsten AF. A role for norepinephrine in stress-induced cognitive deficits: alpha-1-adrenoceptor mediation in the prefrontal cortex. Biol Psychiatry. 1999 Nov 1;46(9):1266-74. doi: 10.1016/s0006-3223(99)00138-9. PMID 10560032
- [Background] Hieble JP, Ruffolo RR Jr. The use of alpha-adrenoceptor antagonists in the pharmacological management of benign prostatic hypertrophy: an overview. Pharmacol Res. 1996 Mar;33(3):145-60. doi: 10.1006/phrs.1996.0022. PMID 8880886
- [Background] Skelly MJ, Weiner JL. Chronic treatment with prazosin or duloxetine lessens concurrent anxiety-like behavior and alcohol intake: evidence of disrupted noradrenergic signaling in anxiety-related alcohol use. Brain Behav. 2014 Jul;4(4):468-83. doi: 10.1002/brb3.230. Epub 2014 Apr 14. PMID 25161814
- [Background] Pickworth WB, Sharpe LG, Nozaki M, Martin WR. Sleep suppression induced by intravenous and intraventricular infusions of methoxamine in the dog. Exp Neurol. 1977 Dec;57(3):999-1011. doi: 10.1016/0014-4886(77)90123-6. No abstract available. PMID 923685
- [Background] Boynton L, Bentley J, Strachan E, Barbato A, Raskind M. Preliminary findings concerning the use of prazosin for the treatment of posttraumatic nightmares in a refugee population. J Psychiatr Pract. 2009 Nov;15(6):454-9. doi: 10.1097/01.pra.0000364287.63210.92. PMID 19934720
- [Background] Raskind MA, Peskind ER, Kanter ED, Petrie EC, Radant A, Thompson CE, Dobie DJ, Hoff D, Rein RJ, Straits-Troster K, Thomas RG, McFall MM. Reduction of nightmares and other PTSD symptoms in combat veterans by prazosin: a placebo-controlled study. Am J Psychiatry. 2003 Feb;160(2):371-3. doi: 10.1176/appi.ajp.160.2.371. PMID 12562588
- [Background] Raskind MA, Peterson K, Williams T, Hoff DJ, Hart K, Holmes H, Homas D, Hill J, Daniels C, Calohan J, Millard SP, Rohde K, O'Connell J, Pritzl D, Feiszli K, Petrie EC, Gross C, Mayer CL, Freed MC, Engel C, Peskind ER. A trial of prazosin for combat trauma PTSD with nightmares in active-duty soldiers returned from Iraq and Afghanistan. Am J Psychiatry. 2013 Sep;170(9):1003-10. doi: 10.1176/appi.ajp.2013.12081133. PMID 23846759
- [Background] George KC, Kebejian L, Ruth LJ, Miller CW, Himelhoch S. Meta-analysis of the efficacy and safety of prazosin versus placebo for the treatment of nightmares and sleep disturbances in adults with posttraumatic stress disorder. J Trauma Dissociation. 2016 Jul-Sep;17(4):494-510. doi: 10.1080/15299732.2016.1141150. Epub 2016 Feb 2. PMID 26835889
- [Background] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655
- [Background] Simpson TL, Malte CA, Dietel B, Tell D, Pocock I, Lyons R, Varon D, Raskind M, Saxon AJ. A pilot trial of prazosin, an alpha-1 adrenergic antagonist, for comorbid alcohol dependence and posttraumatic stress disorder. Alcohol Clin Exp Res. 2015 May;39(5):808-17. doi: 10.1111/acer.12703. Epub 2015 Apr 1. PMID 25827659
- [Background] Rodgman C, Verrico CD, Holst M, Thompson-Lake D, Haile CN, De La Garza R 2nd, Raskind MA, Newton TF. Doxazosin XL reduces symptoms of posttraumatic stress disorder in veterans with PTSD: a pilot clinical trial. J Clin Psychiatry. 2016 May;77(5):e561-5. doi: 10.4088/JCP.14m09681. PMID 27249080
- [Background] Issa SA, Hadid OH, Baylis O, Dayan M. Alpha antagonists and intraoperative floppy iris syndrome: A spectrum. Clin Ophthalmol. 2008 Dec;2(4):735-41. doi: 10.2147/opth.s2697. PMID 19668424
- [Background] Ruiz MA, Zamorano E, Garcia-Campayo J, Pardo A, Freire O, Rejas J. Validity of the GAD-7 scale as an outcome measure of disability in patients with generalized anxiety disorders in primary care. J Affect Disord. 2011 Feb;128(3):277-86. doi: 10.1016/j.jad.2010.07.010. Epub 2010 Aug 9. PMID 20692043
- [Background] Zaider TI, Heimberg RG, Fresco DM, Schneier FR, Liebowitz MR. Evaluation of the clinical global impression scale among individuals with social anxiety disorder. Psychol Med. 2003 May;33(4):611-22. doi: 10.1017/s0033291703007414. PMID 12785463
- [Background] Carlozzi NE, Kratz AL, Downing NR, Goodnight S, Miner JA, Migliore N, Paulsen JS. Validity of the 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) in individuals with Huntington disease (HD). Qual Life Res. 2015 Aug;24(8):1963-71. doi: 10.1007/s11136-015-0930-x. Epub 2015 Jan 31. PMID 25636661
- [Background] Clarke DE, Kuhl EA. DSM-5 cross-cutting symptom measures: a step towards the future of psychiatric care? World Psychiatry. 2014 Oct;13(3):314-6. doi: 10.1002/wps.20154. No abstract available. PMID 25273306
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Zuithoff NP, Vergouwe Y, King M, Nazareth I, van Wezep MJ, Moons KG, Geerlings MI. The Patient Health Questionnaire-9 for detection of major depressive disorder in primary care: consequences of current thresholds in a crosssectional study. BMC Fam Pract. 2010 Dec 13;11:98. doi: 10.1186/1471-2296-11-98. PMID 21144018
- [Background] Maier W, Buller R, Philipp M, Heuser I. The Hamilton Anxiety Scale: reliability, validity and sensitivity to change in anxiety and depressive disorders. J Affect Disord. 1988 Jan-Feb;14(1):61-8. doi: 10.1016/0165-0327(88)90072-9. PMID 2963053
- [Background] Raskind MA, Peskind ER, Chow B, Harris C, Davis-Karim A, Holmes HA, Hart KL, McFall M, Mellman TA, Reist C, Romesser J, Rosenheck R, Shih MC, Stein MB, Swift R, Gleason T, Lu Y, Huang GD. Trial of Prazosin for Post-Traumatic Stress Disorder in Military Veterans. N Engl J Med. 2018 Feb 8;378(6):507-517. doi: 10.1056/NEJMoa1507598. PMID 29414272